CLINICAL TRIAL: NCT06398483
Title: Comparative Study Between Micro Plate Fixation and Blocking k.Wire in Management of Acute Bony Mallet Finger : Randomized Controlled Clinical Trial Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Mohamed Elsadik, Resident at orthopedics and trauma surgery department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-04-06MS
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Bony Mallet Finger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A : acute bony mallet finger managed by micro plate fixation
  Interventions: Procedure: surgical fixation of acute bony mallet finger
- Group B (Active Comparator): Group B : Acute bony mallet finger managed by blocking k.wire fixation
  Interventions: Procedure: surgical fixation of acute bony mallet finger

INTERVENTIONS:
Procedure: surgical fixation of acute bony mallet finger — surgical fixation of acute bony mallet finger by micro plate will be performed under either Infraclavicular nerve blockage or digital block will be performed in all patients .fracture fragment will be reduced, The legs of the plate will be embedded in the terminal tendon to grasp the fragment. The plate will be fixed to the distal phalanx with a 1.3-mm screw.
  surgical fixation of acute bony mallet finger by blocking K.wire will be performed under either infraclavicular nerve block or digital block. The injury will be surgically intervened with an extensor blocking k.wire. the distal phalanx was extended to maximum flexion and (K.wire) will be placed in the cephalic direction through the terminal band at an angle of 45 degrees to the mid-phalanx. Reduction of the fracture fragment will be achieved by bringing the distal phalanx to extension . the DIP will be transfixed with a second K-wire

SUMMARY:
Mallet finger is an avulsion fracture of the distal phalanx or rupture of the extensor terminal band caused by distal interphalangeal (DIP) joint hyperflexion or axial loading. In the treatment of mallet finger fractures, surgical repair is recommended in cases where the fracture involves more than one-third of the distal phalanx joint surface or the distal phalanx becomes volar subluxated

The blocking k.wire and micro plate technique are some of the methods used in the treatment of mallet finger fractures In recent years, the blocking k.wire technique has gained popularity owing to its minimally invasive nature and its ability to achieve satisfactory postoperative results

The main advantages of Micro Plate technique include provision of anatomical reduction and stable fixation, avoiding the risk of fragmentation of the small dorsal fragment, allowing early movement and increasing patient comfort and compliance

ELIGIBILITY:
Inclusion Criteria:

- Acute bony mallet finger involves more than one third of the distal phalanx joint surface or the distal phalanx becomes volar sublaxed

Exclusion Criteria:

1- . crushed distal phalanx 2. soft tissue mallet 3. multiple phalangeal fractures 4. old neglected cases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
post operative evalution of management of acute bony mallet finger | 6 months
  Clinical evaluation of improvement of pain , deformity , range of motion , incidence of surgical site infection , radiographic union time

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided